CLINICAL TRIAL: NCT05820555
Title: Experimental Effects of Children's Evening Media Use on Circadian Phase, Sleep and Executive Functioning
Brief Title: The Goodnight Screen Media Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); William Marsh Rice University (Other); University of Nevada, Reno (Other)
Responsible Party: Principal Investigator, Jennette P. Moreno, PhD, Assistant Professor, Pediatrics - Nutrition, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H-52269; P01 HD109876-01 5256 (Other Grant/Funding Number: NICHD); P01HD109876-01 (NIH)
Record Dates: First submitted 2023-02-13; First posted 2023-04-19 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Sleep; Sleep Hygiene
Keywords: circadian phase; sleep; evening screen media use
MeSH Terms: conditions — Sleep Hygiene

STUDY DESIGN:
Intervention Model Description: A 3-group randomized controlled trial design will be used in which children are assigned to receive one of 2 experimental conditions or a control condition
Who Masked: Investigator
Masking Description: Blinding of the study biostatistician and PI during the analysis will be ensured. Groups will be denoted by a variable that does not reveal its identity. The blinding will be broken after the data set is closed and analyses completed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A: 1 hour of tablet use in the hour before bed (Experimental): During week 1, children will maintain a sleep schedule within 30 minutes +/- of their habitual bedtime. This bedtime will be maintained throughout the 3 weeks of the study except on nights when dim light melatonin onset is assessed in the lab.
  During week 2, participants will be asked to reframe from screen use in the 3 hours before bed time for 6 evenings.
  During week 3, participants will be exposed to 1 hour of tablet use (Standard bright setting), 1 hour before bedtime for 6 evenings.
  Interventions: Behavioral: Timed evening technology and digital media use (tablet use)
- Group B: 1 hour of tablet use 2 hours before bed (Experimental): During week 1, children will maintain a sleep schedule within 30 minutes +/- of their habitual bedtime. This bedtime will be maintained throughout the 3 weeks of the study except on nights when dim light melatonin onset is assessed in the lab.
  During week 2, participants will be asked to reframe from screen use in the 3 hours before bedtime for 6 evenings.
  During week 3, participants will be exposed to 1 hour of tablet use (Standard bright setting), 2 hours before bedtime (and no screen use in the hour before bed) for 6 evenings.
  Interventions: Behavioral: Timed evening technology and digital media use (tablet use)
- Control Condition (Active Comparator): During week 1, children will maintain a sleep schedule within 30 minutes +/- of their habitual bedtime. This bedtime will be maintained throughout the 3 weeks of the study except on nights when dim light melatonin onset is assessed in the lab.
  During week 2, participants will engage no screen use for the 3 hours before bedtime for 6 evenings.
  During week 3, participants will be asked to engage in no screen use in the 3 hours before bedtime for 6 evenings.
  Interventions: Behavioral: no technology and digital media use (screen media use)

INTERVENTIONS:
Behavioral: Timed evening technology and digital media use (tablet use) — timing of children's evening tablet device use relative to bedtime
  Arms: Group A: 1 hour of tablet use in the hour before bed; Group B: 1 hour of tablet use 2 hours before bed
Behavioral: no technology and digital media use (screen media use) — no screen media use relative to bedtime (Tablets, computers, TV, moble devices, smart phone)
  Arms: Control Condition

SUMMARY:
To test the timing of evening tablet use on children's circadian phase and sleep (i.e., sleep onset and sleep duration) compared to no screen media use. To explore the effect of evening tablet use on children's inhibitory control and executive function.

DETAILED DESCRIPTION:
The goal of the study is to test the effect of tablet use before bed on the sleep, circadian phase, and executive functioning (EF) of 4-year-olds using a 3-group randomized controlled trial in which children are assigned to receive one of 2 experimental conditions (Group A:1 hour of tablet use in the hour before bed; Group B:1 hour of tablet use 2 hours before bed) or a control condition (no evening screen media use). It is hypothesized that in comparison to no tablet use, daily exposure to tablet use before bed will be associated with a delay in children's circadian phase (e.g., occurring later in the evening/night), a longer sleep latency (i.e., later sleep onset), and shorter sleep duration. It is anticipated that tablet use in the hour before bed will have a greater impact on children's circadian phase and sleep than tablet use 2 hours before bed, or no tablet use before bed. We will explore whether changes in circadian phase and sleep result in poorer performance on measures of EF (i.e., inhibitory control and working memory).

ELIGIBILITY:
Inclusion Criteria:

* preschool-aged children (4.0 to <5.0 years old) and their parent
* living in the Greater Houston area.
* parent must be a biological parent or legal guardian who lives with the child ≥50% of the time and has a primary role of caring for the child
* parent is comfortable participating in the study and responding to questionnaires in English.
* The child does not have to have access to mobile device, but if they do, the primary device they use has to be an Android OS ≥5.0 either used only by the study child or shared with others, or an Apple iOS ≥14.0 that only the child uses.
* Parent and child must be fluent in English.

Exclusion Criteria:

* The child has a chronic medical condition or takes a medication affecting sleep, or circadian rhythms (e.g., melatonin supplementation, diagnosed sleep disorder, steroid use, etc.) or a diagnosed cognitive or learning impairment affecting EF (e.g., attention deficit hyperactivity disorder).
* Child with blindness or significant vision problems that impacts both screen media use and sleep.

Ages: 48 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2023-04-24 (Actual); Primary Completion 2026-05-28 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Dim light Melatonin Onset Phase | Day 7 to Day 14
  Circadian phase can be examined by measuring the circadian timing of melatonin onset under dim light conditions (dim light melatonin onset; DMLO). Compared to markers of endogenous circadian rhythms, melatonin is relatively robust. Salivary DLMO measures have demonstrated high intraclass correlations (.93) with plasma and sensitivity and specificity comparable to plasma assays. Following established procedures with children, salivary DLMO will be collected on a in the laboratory under dim light conditions (<5 lux), via a cheek swab every 30-60 minutes beginning 5 hours prior to and ending 1-hour following typical bedtime. Saliva samples will be centrifuged, frozen, and assayed using radioimmunoassay test kits by Solid Phase in Portland Me. DLMO phase will be determined using linear interpolation across the time points before and after melatonin concentration increased to and remained above 4pg/mL.
Change in Dim light Melatonin Onset Phase | Day 14 to Day 21
  Circadian phase can be examined by measuring the circadian timing of melatonin onset under dim light conditions (dim light melatonin onset; DMLO). Compared to markers of endogenous circadian rhythms, melatonin is relatively robust. Salivary DLMO measures have demonstrated high intraclass correlations (.93) with plasma and sensitivity and specificity comparable to plasma assays. Following established procedures with children, salivary DLMO will be collected on a in the laboratory under dim light conditions (<5 lux), via a cheek swab every 30-60 minutes beginning 5 hours prior to and ending 1-hour following typical bedtime. Saliva samples will be centrifuged, frozen, and assayed using radioimmunoassay test kits by Solid Phase in Portland Me. DLMO phase will be determined using linear interpolation across the time points before and after melatonin concentration increased to and remained above 4pg/mL.

SECONDARY OUTCOMES:
Change in the Average Sleep Onset | Day 1 through 6 to Day 9 through Day 13
  Actigraphs (GT3X-BT, Pensacola, FL) worn on the wrist of the non dominant hand 24 hours a day for 4-5 days will measure sleep duration and timing of sleep onset and waking. Wrist placement reliably measures sleep duration. Sleep diaries will be completed. Monitor-wear logs will identify times the accelerometer is removed and the activity engaged in while the monitor is off.
Change in the Average Sleep Onset | Day 9 through 13 and Day 16 through 20
  Actigraphs (GT3X-BT, Pensacola, FL) worn on the wrist of the non dominant hand 24 hours a day for 4-5 days will measure sleep duration and timing of sleep onset and waking. Wrist placement reliably measures sleep duration. Sleep diaries will be completed. Monitor-wear logs will identify times the accelerometer is removed and the activity engaged in while the monitor is off.
Change in Average Sleep duration | Day 1 through 6 to Day 9 through Day 13
  Actigraphs (GT3X-BT, Pensacola, FL) worn on the wrist of the non dominant hand 24 hours a day for 4-5 days will measure sleep duration and timing of sleep onset and waking. Wrist placement reliably measures sleep duration. Sleep diaries will be completed. Monitor-wear logs will identify times the accelerometer is removed and the activity engaged in while the monitor is off.
Change in Average Sleep duration | Day 9-13 and Day 16-20
  Actigraphs (GT3X-BT, Pensacola, FL) worn on the wrist of the non dominant hand 24 hours a day for 4-5 days will measure sleep duration and timing of sleep onset and waking. Wrist placement reliably measures sleep duration. Sleep diaries will be completed. Monitor-wear logs will identify times the accelerometer is removed and the activity engaged in while the monitor is off.
Change in Inhibitory Control-Day/Night | Day 14 or Day 21
  Children's inhibitory control will be assessed using the Day/Night task. The order of this task will be counterbalanced across Day 14 and 21. This task can be used interchangeably with Grass/snow, so we will examine the difference in performance from the test administered on day 14 to the test administered on day 21.
Change in Inhibitory Control-Grass/Snow | Day 14 or Day 21
  Children's inhibitory control will be assessed using the Grass/Snow. The order of this task will be counterbalanced across Day 14 and 21. This task can be used interchangeably with Grass/snow, so we will examine the difference in performance from the test administered on day 14 to the test administered on day 21.
Change in Working memory | Day 14 to Day 21
  Children's Working Memory will be assessed using the Missing Scan assessment. This task will be administered at Day 14 and 21.
Change in Working memory | Day 14 to Day 21
  Children's Working Memory will be assessed using the Spin the Pots assessment. This task will be administered at Day 14 and 21.
Change in combined assessment of Executive Functioning working memory and inhibitory control | Day 14 to Day 21
  The Head-Toes-Knees-Shoulder Task assesses both working memory and inhibitory control and will be administered on Day 14 and Day 21.

OTHER OUTCOMES:
Ambient Light Exposure | Days 1-21
  ActLumus devices containing a photocell will be used to assess ambient light exposure. Devices will be pinned to the shirt. ActLumus devices are capable of assessing light intensity and wavelength. Light exposure will be used as a covariate in analyses.
Average daily duration of Tablet use (excluding the experimental exposures) | Days 1-21
  Children's tablet use on Android and iOS devices will be assessed during the study period. Daily screen use will be used as a covariate in the analysis. The Chronicle app will be used to assess the timing and amount of children's Android device use. Code developed by Arcascope will be used to assess the amount of children's iOS device usage.
Percentage of time that children followed the screen media use guidelines for their condition during week 2 | Days 8-13
  The Chronicle and Acrascope data will be used to assess adherence to the evening tablet use conditions.
Percentage of time that children followed the screen media use guidelines for their condition during week 3 | Days 15-20
  The Chronicle and Acrascope data will be used to assess adherence to the evening tablet use conditions.
Children's Sleep Hygiene Scale (total score) | Day 7
  Sleep hygiene will be assessed by parent report on the Children's Sleep Hygiene Scale. Contains 22 items. Response options are scored as follows: Never (1 point); Once in Awhile (2 points); Sometimes (3 points); Quite Often (4 points); Frequently, if not Always (5 points); Always (6 points). It contains 6 subscales that are computed by computing the mean of the items (each subscale could range from 1-6). The total score is computed by computing the mean of the subscales, with a potential range of 1-6. The total score will be used as the outcome of interest in the current study. Higher scores indicate better sleep hygiene practices.
The Children's Chronotype Questionnaire | Day 7
  Chronotype will be assessed by parent report of the child's preference for morningness or eveningness. The M/E score is calculated by adding items 17-26 (responses scored as a=1, b=2, c=3, d=4, d=5), except items 17,18,24,25 are reverse scored. the M/E score ranges from 10 (extreme morningness) to 49 (extreme eveningness). Morning types are defined as having a M/E scale score of ≤23, intermediate types: score of 24-32, and evening types: score ≥33.
Children's Sleep Habits Questionnaire | Day 7
  Parents will be asked to report children's sleep behaviors and problems on the Child Sleep Habits Questionnaire. The total sleep disturbance score is comprised of 33 items. Response options are scored as Usually = 3; Sometimes = 2; and Never/Rarely = 1. Scores range from 33 to 99. Higher scores indicate more sleep problems.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Nutrition Research Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
The principal investigator and co-investigators acknowledge their willingness to share data with other eligible investigators through academically established means. Summarized data will be shared with collaborators as soon as available, with local colleagues at seminars and talks, and with the scientific community at large by posters and presentations at local, regional, national and international scientific meetings.
  Individual participant data may be shared in accordance with the NIH data sharing policy.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: All de-identified scientific data generated by the study, and any necessary metadata (including, but not limited to, study protocols and documentation on data collection instruments), will be deposited in the NICHD-maintained Data and Specimen Hub (DASH) data repository no later than at the time of acceptance for an associated publication, or at the end of funding period, whichever is sooner.
  Code will be shared via the Rice team's webpage at https://computationalimaging.rice.edu/code/ or via GitHub
Access Criteria: Users of the DASH repository must agree to the DASH user agreement
URL: https://dash.nichd.nih.gov/